CLINICAL TRIAL: NCT03452202
Title: Using tDCS in Speech-based Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-01474
Record Dates: First submitted 2018-01-16; First posted 2018-03-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Apraxia of Speech
Keywords: Stroke
MeSH Terms: conditions — Apraxias; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Stimulation (Experimental): crossover design such that each participant receives behavioral treatment twice - once with active stimulation and once with sham stimulation - in order to evaluate differences in improvement based on treatment condition.
  Interventions: Device: Soterix 1x1 line tDCS low-intensity stimulator; Device: Sham
- Sham Stimulation (Sham Comparator): crossover design such that each participant receives behavioral treatment twice - once with active stimulation and once with sham stimulation - in order to evaluate differences in improvement based on treatment condition.
  Interventions: Device: Soterix 1x1 line tDCS low-intensity stimulator; Device: Sham

INTERVENTIONS:
Device: Soterix 1x1 line tDCS low-intensity stimulator — Introduction of the independent variable (treatment) across three different points in time. Participants will be randomly assigned to have each treatment phase begin after 3, 4, or 6 baseline sessions. This current stimulates the cortex, with anodal stimulation leading to a depolarized state in which neurons are more likely to fire.
  Other Names: Soterix
Device: Sham — Patients will have two electrodes applied (one anode, one cathode) administering no stimulation

SUMMARY:
The purpose of this study is to determine whether the effect of treatment for acquired speech impairment can be enhanced by combining effective behavioral treatment with non-invasive brain stimulation. Transcranial direct current stimulation (tDCS), which delivers low-intensity current to the scalp, and is a safe and well-tolerated approach that poses a non-significant risk to participants. tDCS provides low intensity neural stimulation which has been shown to facilitate motor learning in other domains of stroke rehabilitation such as arm motor learning but the potential to enhance speech motor learning has not been explored. This will be examined with a series of single-case experimental designs.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Monolingual (English)
* Single left-hemisphere CVA
* A minimum of six months post-stroke
* Clinical diagnosis of apraxia of speech
* Normal speech perception
* Passing score on the hearing screening.

Exclusion Criteria:

* Diagnosis of laryngeal voice disorder
* Dysarthria
* History of speech impairment prior to CVA
* Presence of potential tDCS risk factors: damaged skin at site of stimulation;
* Presence of electrically or magnetically activated implant (including pacemaker);
* metal in any part of their body;
* history of medication-resistant epilepsy in the family;
* past history of seizures or unexplained spells of loss of consciousness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in accuracy in recordings from tasks from baseline to post treatment | Baseline, 6 Months
  Subjects will be given speech production tasks. Recordings of tasks will be scored for accuracy to measure speech motor learning

CONTACTS AND LOCATIONS:
Overall Officials: Adam Buchwald, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - Burke Rehabilitation Hospital, White Plains, New York